CLINICAL TRIAL: NCT02536729
Title: Evaluation of the Quality of Life of Patients Requiring Intestinal Cleansing Using Oral Medications to Imaging Procedure by Patient Reported Outcome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fundación Salutia (Other)
Collaborators: Tecnoquimicas S.A (Unknown)
Responsible Party: Sponsor
Other Study IDs: TRAVAD2015
Record Dates: First submitted 2015-08-27; First posted 2015-09-01 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Bowel Preparation
MeSH Terms: interventions — Polyethylene Glycols; Electrolytes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Oral Sodium Phosphate - Normal preparation: Oral sodium phospate exposure with special diet (Liquid)
  Interventions: Drug: Oral Sodium Phosphate - Normal preparation
- Oral Sodium Phosphate - Modified preparation: Oral sodium phospate exposure with special diet (Liquid), but the participant can normally lunch the day before the test
  Interventions: Drug: Oral sodium phosphate - Modified Preparation
- polyethylene glycol + Electrolytes: polyethylene glycol + Electrolytes exosure with special diet (Liquid)
  Interventions: Drug: polyethylene glycol + Electrolytes

INTERVENTIONS:
Drug: Oral Sodium Phosphate - Normal preparation
  Other Names: Travad
  Groups: Oral Sodium Phosphate - Normal preparation
Drug: Oral sodium phosphate - Modified Preparation
  Other Names: Travad
  Groups: Oral Sodium Phosphate - Modified preparation
Drug: polyethylene glycol + Electrolytes
  Other Names: PEG
  Groups: polyethylene glycol + Electrolytes

SUMMARY:
Objective: The primary objective of this study is to assess the quality of life of people treated with oral phosphate compared with polyethylene glycol + electrolytes to imaging procedures, according to the outcome variables reported by patients.

Type of study: A non-interventional observational analytic prospective cohort study.

Sample: We will include people who need bowel cleansing for the realization of imaging tests

Exposures: - oral sodium phosphate normal regimen

* Oral sodium phosphate with modified diet
* Polyethylene Glycol + electrolytes

Follow-up time: 8 days after the bowel preparation

Outcomes: Boston Scale measure Safety Differences between groups in blood test (Sodium, Potassium, Calcium)

ELIGIBILITY:
Inclusion Criteria:

* Patients which have order for an imaging procedure that requires bowel cleansing
* Older than 18 years and younger than 65 years old
* Accept to participate in this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults who are in diagnostic centers, which have order for an imaging procedure that requires intestinal cleansing conducted.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Boston scale for bowel cleansing | 2 days

SECONDARY OUTCOMES:
Number of adverse events | 8 days
Quality of life | 8 days
  Quality of life measured with EQ5D-3L scale
Blood creatinine | 8 days
Blood urea nitrogen (BUN) | 8 days
Blood Sodium | 8 days
Blood Potassium | 8 days
Blood Calcium | 8 days
Blood Phosphorus | 8 days